CLINICAL TRIAL: NCT06845982
Title: Anatomopathological Evaluation of a New Ultrasound-guided Transuterine Vaginal Biopsy Technique in Uterine Fibromatous Disease
Acronym: EFIBIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RCAPHM23_0387; 2024-A01337-40 (Other: RCB)
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Uterine Fibroids (UF)
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ultrasound-guided transuterine vaginal biopsy (BVTE) (Experimental): A BVTE is performed under general anaesthetic in the operating theatre on the scheduled day of myomectomy or hysterectomy. It will be directed to the centre of the uterine smooth muscle tumour in question via an exclusively transuterine route to avoid any peritoneal spread. At least 4 to 5 samples will be taken per uterine smooth muscle tumour, with a maximum of 3 tumours to limit the risk of confusion. The woman will then be operated on as planned during the same operation. All surgical specimens will be sent to the Anatomopathology Department of La Timone for anatomopathological diagnosis after immediate formalin embedding during surgery. Surgical specimens will be analysed as usual.
  Interventions: Other: ultrasound-guided transuterine vaginal biopsy (BVTE)

INTERVENTIONS:
Other: ultrasound-guided transuterine vaginal biopsy (BVTE) — A BVTE is performed under general anaesthetic in the operating theatre on the scheduled day of myomectomy or hysterectomy. It will be directed to the centre of the uterine smooth muscle tumour in question via an exclusively transuterine route to avoid any peritoneal spread. At least 4 to 5 samples will be taken per uterine smooth muscle tumour, with a maximum of 3 tumours to limit the risk of confusion. The woman will then be operated on as planned during the same operation. All surgical specimens will be sent to the Anatomopathology Department of La Timone for anatomopathological diagnosis after immediate formalin embedding during surgery. Surgical specimens will be analysed as usual.

SUMMARY:
The benign uterine fibroid is part of the broader term uterine smooth muscle tumour, which also includes malignant myometrial tumours (MSTs) of varying malignancy (uterine sarcoma, cellular fibroid, STUMP (uterine smooth muscle tumours of uncertain malignant potential)).

Magnetic resonance imaging (MRI) is the most effective test for distinguishing a fibroid from a TMM, but its reliability is limited. This leads to inappropriate management in a number of situations. The first is the risk of overtreatment by performing surgery for a suspected TMM on MRI in a patient with few or no symptoms and a final histological diagnosis of fibroid. The second is the risk of unsatisfactory or even harmful cancer surgical treatment in a symptomatic patient with a reassuring MRI diagnosis but a final histological diagnosis of TMM. Finally, there is the possibility of treating a lesion labelled as a fibroid on MRI with an alternative technique (embolisation, radiofrequency, HIFU) when it is in fact a TMM, thereby delaying appropriate treatment and worsening the prognosis.

Ultrasound-guided transuterine vaginal biopsy (ETVB) is an innovative and promising minimally invasive technique for preoperative anatomopathological diagnosis. It would make it possible to obtain a histological diagnosis without the need for surgery, thereby avoiding the inappropriate management described above.

The aim of this study is to validate an innovative minimally invasive surgical technique (BVTE) for the diagnosis of uterine smooth muscle tumours by biopsy, to assess the complications associated with the technique and any potential adverse effects, and to evaluate the feasibility of the technique in current practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age consulting the CHU de la Conception who require surgical treatment for uterine smooth muscle tumours (fibroma or TMM).
* Able to give written consent
* Beneficiary or beneficiary of a social security scheme

Exclusion Criteria:

* Person in a period of exclusion from another research protocol at the time of signing consent/no objection
* Subjects covered by articles L1121-5 to 1121-8 of the Public Health Code, i.e. :
* Pregnant women, women in labour and nursing mothers
* Persons deprived of their liberty by judicial or administrative decision
* Persons subject to psychiatric monitoring under articles L3112-1 and L3113-1 who are not covered by the provisions of article L1121-8
* Minors
* Adults subject to a legal protection measure or unable to express their consent.
* A person who does not have a sufficient command of reading and understanding the French language to be able to consent to participate in the research.
* Any other reason which, in the opinion of the investigator, could compromise the safety of the research participant and/or interfere with the evaluation of the objectives of the research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Anatomopathological analysis of biopsy with BVTE technique and comparison with the reference technique | Form enrollement to the end of the study at 43 months
  The main aim of our study will be to evaluate the diagnostic performance of a BVTE biopsy technique for preoperative uterine smooth muscle tumours to discriminate between fibroids and MCTs.

SECONDARY OUTCOMES:
Number of intraoperative complications according to the Clavien-Dindo classification | During the surgery
  The secondary objective of this study will be to count the numbre of intraoperatoire complications associated with the BVTE technique, in comparison with the reference technique.
Number of postoperative complications according to the Clavien-Dindo classification | From the surgery to the end of the study at 43 months
  The secondary objective of this study will be to count the numbre of postoperatoire complications associated with the BVTE technique, in comparison with the reference technique.

OTHER OUTCOMES:
Number of equipment in accordance with number of patients in current practice | From enrollement to the end of the study at 43 months
  The exploratory objectives will be to assess the feasibility of the technique in current practice. So investigators will evaluate the number of equipment available for the technique in current practice in comparison with a reference technique.
Cost (euros) of the BVTE technique in current practice | From enrollement to the end of the study at 43 months
  The exploratory objectives will be to assess the feasibility of the technique in current practice. So investigators will evaluate the cost of the technique in current practice in comparison with a reference technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Conception, Marseille, France